CLINICAL TRIAL: NCT02789852
Title: Evaluation of the Effectiveness of Night Orthosis in Treating Women With Symptomatic Osteoarthritis in the Interphalangeal Joint of the Dominant Hand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Paula Gabriel Silva, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PGSilva
Record Dates: First submitted 2016-05-23; First posted 2016-06-03 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Hand Injuries
MeSH Terms: conditions — Hand Injuries | interventions — Orthotic Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Orthosis Group (Experimental): Will use the night orthosis for interphalangeal in the treatment of OA hand.
  Interventions: Device: Orthosis
- Control Group (No Intervention): wait for treatment

INTERVENTIONS:
Device: Orthosis — use orthosis
  Arms: Orthosis Group

SUMMARY:
Evaluation of the effectiveness of using a night orthosis for II and III or fingers of the dominant hand in women diagnosed with symptomatic osteoarthritis compared to a control group.

DETAILED DESCRIPTION:
Objective: To evaluate the effectiveness of using a night orthosis for II and III or fingers of the dominant hand in women diagnosed with symptomatic osteoarthritis compared to a control group.

Methods: Through a randomized controlled clinical trial with blind assessment and follow-up of six months. Fifty-Two participants were randomized into two groups: group orthosis and control, and made a night orthosis II and or III fingers, thermoplastic will be used as a treatment for participants orthosis group. The participants underwent four evaluations at time 0, 45 days, 90 days and 180 days after its inclusion in the study. The variables studied were: the visual analog scale of pain, grip and pinch strength, questionnaires Cochin and Australian/Canadian Hand Osteoarthritis Index and functional Pick-up test.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 40 and 80 years.
* Patients diagnosed with osteoarthritis (OA) hand according to the American College of Rheumatology classification criteria.
* Pain symptom in proximal interphalangeal (PIP's) or distal interphalangeal (DIP's) dominant hand in II and III or fingers.
* Provide greater pain symptom of II and III or fingers between each other.
* Complains of pain symptom measured by a visual analog scale (VAS) pain between 3 to 8 cm in the II and III or fingers of the dominant hand reported to perform joint movement (activity).
* Thumb abduction with the II and III fingers without changing the pincer movement pulp-pulp.

Exclusion Criteria:

* Other rheumatic diseases, neurological and skeletal muscle that can affect the upper limb.
* Fibromyalgia uncontrolled.
* Pregnancy.
* Geographical inaccessibility and transport.
* Cognitive impairment that prevents the understanding of assessment tools.

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in Pain | T0 (inclusion), T45( 45 days after inclusion), T90 (90 days after inclusion) and T180 (180 days after inclusion)
  Pain was assessed using the visual analog scale ranging from 0 cm to 10 cm

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Sao Paulo, São Paulo, São Paulo, Brazil